CLINICAL TRIAL: NCT01523353
Title: Feasibility Study of Preoperative Exercise Intervention in the Resection of Colorectal Liver Metastasis.
Brief Title: Prehabilitation in Liver Surgery
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Liverpool University Hospitals NHS Foundation Trust (Other Government)
Responsible Party: Principal Investigator, Declan Dunne, Surgical Research Fellow, Liverpool University Hospitals NHS Foundation Trust
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 11/H1005/3
Record Dates: First submitted 2012-01-30; First posted 2012-02-01 (Estimated); Last update posted 2013-12-17 (Estimated); Status verified 2012-02

CONDITIONS: Colorectal Cancer; Colorectal Liver Metastasis; Liver Surgery; Exercise Intervention
Keywords: Prehabilitation; Exercise; Colorectal Cancer; Surgery
MeSH Terms: conditions — Colorectal Neoplasms; Motor Activity

STUDY DESIGN:
Who Masked: Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Exercise Intervention (Active Comparator): 4 week personalised exercise program on a static bicycle.
  Interventions: Behavioral: Exercise Intervention
- Control Arm (No Intervention): Patients having standard preoperative preparation and advice.

INTERVENTIONS:
Behavioral: Exercise Intervention — 4 week personalised exercise program on a static cycle. Supervised in a hospital environment
  Arms: Exercise Intervention

SUMMARY:
Each year in the UK around 1500 patients undergo surgery for bowel cancer that has spread to the liver. This is major surgery that offers a chance of cure, but can be associated with complications. Fitter patients are less likely to have serious complications. We are interested in finding out whether a short exercise program can improve patient fitness before surgery and whether this can reduce surgical complications.

We plan to measure the fitness of patients who are going to have liver surgery. We will then give them an exercise programme for 4 weeks, after which we will assess their fitness again.

We are also interested in whether fitter people have better Liver function. To assess this we will take a small sample of liver tissue during the operation for laboratory analysis of its function.

Hypothesis

1. A short period of exercise can significantly improve fitness prior to liver surgery
2. Greater Fitness is associated with better liver function.

DETAILED DESCRIPTION:
Prehabilitation in Liver Surgery

Introduction Thirty per cent of patients with colorectal cancer have metastatic disease at time of presentation, and a further 20% will develop liver metastases after the primary colorectal malignancy has been resected. Liver resection offers the prospect of cure for a proportion of these patients and, with the increasing use of effective neo-adjuvant chemotherapy, this proportion is increasing. However, liver surgery is associated with significant morbidity and mortality and this may be higher in patients with comorbidity, poor cardiorespiratory fitness and in those who have received neo-adjuvant chemotherapy.

Cardiopulmonary exercise testing (CPET) is a non-invasive assessment of cardiovascular and pulmonary function, which can be quantified by measures such as anaerobic threshold (AT) and VO2peak. The anaerobic threshold is a measure of sustainable exercise, where the VO2peak is a measure of maximal exercise capacity. The AT has been assessed in different surgical groups and has been shown as a useful predictor of postoperative complications and survival. Early work has demonstrated that short periods of preoperative exercise intervention can improve AT and VO2peak. However, no work has to date been undertaken in patients prior to liver surgery.

Hepatic glucose metabolism provides much of the energy requirements of the postoperative period. Work has demonstrated that exercise training increases hepatic glucose production, and that its inhibition has a marked effect on endurance capability. This may be particularly relevant when surgical resections can involve resection of up to 80% of hepatic tissue. However, a link between hepatic gluconeogenic capacity and fitness as assessed by cardiopulmonary exercise testing has not been established.

A demonstrable link between gluconeogenic capacity and cardiopulmonary fitness and an explanation of its underpinning physiology would help explain some of the systemic effects of drug hepatotoxicity. It would also allow development of strategies to improve gluconeogenic capacity that may reduce complications and improve tolerance of many hepatoxic agents such as chemotherapy.

Hypothesis

1. A short exercise program can significantly improve the CPET defined anaerobic threshold prior to liver surgery in a cancer population and this will be associated with reduced post-operative morbidity and mortality.
2. Hepatic gluconeogenic capacity will be associated with cardiopulmonary fitness.
3. Gluconeogenic capacity will be associated with mitochondrial number and quantity of enzymes which are integral to gluconeogenesis such as PEPCK

Methods Patients with colorectal liver metastases suitable for hepatic resection will undergo a baseline CPET and then be randomised to either preoperative exercise intervention or standard care. Patients within the intervention arm will undergo a 4 week exercise program consisting of 3 interval sessions per week on a stationary bike. This will be individually tailored according to their initial exercise test. In the week prior to surgery all patients will then undergo a further CPET. At surgery liver tissue will be taken to determine hepatic gluconeogenic capacity. CPET tests will then be performed where possible in patients at 6 weeks and 3 months following surgery. Post-operative complications (Clavien classification and Postoperative morbidity score (POMS)) and 30 and 90-day mortality will be recorded. Quality of life assessments (EORTC/SF-36) will be taken at recruitment, the week prior to surgery, 6 weeks after surgery and 3 months following surgery.

Laboratory Analysis Hepatic gluconeogenic capacity will be assessed by direct analysis of fresh slices of hepatic tissue taken at the time of surgery. Slices will be taken using the Krumdiek MD6000 tissue slicer. These will be weighed an incubated in a buffer containing lactate. Glucose will be measured using the Glucose Oxidase assay, and calculated per mg wet weight of hepatic tissue. Further analysis of mitochondrial number and ATP production, and enzymatic levels will be conducted following initial results.

Statistical considerations This is a study of a continuous response variable from matched pairs of study subjects and will need 38 patients to detect a true difference 1.5ml/min/kg, with a probability 0.8 and Type I error 0.05). Anticipated recruitment period is 10 months assuming a dropout rate of 20%. Randomisation is by computerised block randomisation, and patients will be stratified by receipt of neo-adjuvant chemotherapy.

ELIGIBILITY:
Inclusion Criteria:

* Planned resection of colorectal liver metastasis
* Able to perform cycle based exercise program
* Age over 18

Exclusion Criteria:

* Unable to consent
* Unable to perform cycle based exercise program
* Age under 18

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 37 (Actual)
Dates: Start 2011-07; Primary Completion 2013-06 (Actual); Study Completion 2013-06 (Actual)

PRIMARY OUTCOMES:
Anaerobic threshold prior to liver resection | 4 weeks
  This is a measure of cardiopulmonary fitness as detected by a cardiopulmonary exercise test.

SECONDARY OUTCOMES:
Hospital Length of stay | 6 weeks
  length of hospital admission from date of surgery
Post operative morbidity | 3 months
  As measured using Clavien classification and postoperative morbidity scores
Quality of Life | 4 months
  SF -36 and EORTC questionaires at 5 weeks, 6 weeks postoperatively, and 3 months postoperatively
Mortality | 30 day and 90 day postoperative
Attendance at exercise sessions | 6 weeks
Serious adverse events within exercise program | 6 weeks
  The investigators are not expecting and serious adverse events during the program.
other measures of cardiopulmonary function | 6 weeks
  Detected by cardiopulmonary exercise prior to surgery.
Recovery of fitness | 6 and 12 weeks post operatively
  recovery of cardiopulmonary exercise test determined fitness post surgery.

CONTACTS AND LOCATIONS:
Overall Officials: Declan FJ Dunne, MBChB(Hons), Principal Investigator — Liverpool University Hospitals NHS Foundation Trust
Locations (1):
- Aintree University Hospital, Liverpool, Merseyside, United Kingdom

REFERENCES:
- [Derived] Dunne DF, Jack S, Jones RP, Jones L, Lythgoe DT, Malik HZ, Poston GJ, Palmer DH, Fenwick SW. Randomized clinical trial of prehabilitation before planned liver resection. Br J Surg. 2016 Apr;103(5):504-12. doi: 10.1002/bjs.10096. Epub 2016 Feb 11. PMID 26864728